CLINICAL TRIAL: NCT02350400
Title: Pilot Study to Assess the Safety and Pharmacokinetics of 70-150μm Drug Eluting Beads Loaded With Irinotecan (DEBIRI) in the Treatment of Hepatic Colorectal Metastases
Brief Title: Pilot Study to Assess the Safety and Pharmacokinetics of 70-150μm Drug Eluting Beads Loaded With Irinotecan (DEBIRI).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Singhealth Foundation (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEBIRI_TKH_01_2012
Record Dates: First submitted 2014-11-26; First posted 2015-01-29 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Drug eluting beads; Irinotecan; Pharmacogenetics; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DEBIRI (Experimental): For unilobar disease, two treatments will be planned, separated by four weeks. For bilobar disease, there will be four treatments planned, alternating between right and left lobe, separated by 2 weeks duration.
  Interventions: Device: DEBIRI

INTERVENTIONS:
Device: DEBIRI — DEBIRI TACE
  Other Names: DC Beads loaded with irinotecan; (Manufacturer- Biocompatibles UK Limited)

SUMMARY:
Background

Hepatic metastases of colorectal cancer (MCC) is quite common and is a major source of morbidity and mortality. There has been evidence to show that hepatic arterial chemoembolisation using DC beads (drug eluting beads, 100-300μm) loaded with irinotecan (DEBIRI) showed improved overall survival when compared to systemic therapy (FOLFIRI), but being larger they have their limitations.

New 70-150μm beads are recently available and currently there is limited data concerning its use. Safety of these beads have not been tested in local patients.

Hypothesis / Aim To study the safety and pharmacokinetics of the smaller 70-150μm DEBIRI in a pilot study of 5 patients. The smaller 70-150μm beads will be able to deliver a more consistent and higher dose to tumoral tissue with a smaller systemic dose. Being smaller and less embolic, it will also be better tolerated. Patients will also be genotyped for their UGT1A1*28 and UGT1A1*6 polymorphism status as the latter genotypes are associated with decreased clearance of irinotecan and SN-38 in Asian patients.

Methods Single centre, pilot study, prospectively recruiting 5 patients with unilobar disease, refractory to systemic chemotherapy

The primary endpoints:

1. establish safety and toxicity profile of the irinotecan loaded DEBIRI beads
2. establish pharmacokinetics and systemic exposure of irinotecan and its active metabolite, SN-38.

The secondary outcome measurements:

1. the incidence and severity of adverse events, liver function parameters and laboratory abnormalities;
2. response rate,
3. progression free survival
4. overall survival

Clinical Significance

This treatment modality has the advantage of directly delivering irinotecan to the liver metastases from colorectal cancer. This local mode of drug delivery may result in a higher intratumoral drug concentration and rapid tumour shrinkage leading to downstaging of the hepatic metastatic lesions. These therapeutic outcomes may also downstage patients to hepatic resection.

DETAILED DESCRIPTION:
1. Recruitment:

   Suitable potential subjects will be identified, namely those who have failed first or second line chemotherapy agents.
2. Liver biopsy Right before the 1st transarterial chemoembolisation procedure, the liver metastases will be biopsied under ultrasound or CT guidance by the IR with a 18G core biopsy needle. Tissue will be sent for histological analysis as well as stored for molecular studies with NCCS.
3. Transarterial chemoembolisation procedure (DEBIRI TACE):

100mg of irinotecan will be loaded into the DEB solution at least 2 hours before the procedure by the pharmacy.

Diagnostic angiography (DSA) will performed under fluoroscopic guidance, most commonly via right groin puncture. Using dedicated catheters, arterial supply of the liver and the tumour involved segments will be determined. A solution of 75-150 μm DEBIRI mixed with non-ionic contrast medium (1:1) will be injected into the artery feeding the metastases.

For unilobar disease, two treatments will be planned, each of them with a maximum of 100mg irinotecan loaded in into the DEB, separated by four weeks. Intravenous fentanyl will be administered for procedural pain relief. Post procedural pain relief medications will be given as deemed necessary by the physician.

For bilobar disease, there will be four treatments planned, alternating between the right and left lobe, separated by 2 weeks duration, each of them with a maximum of 100mg irinotecan loaded into the DEB. Intravenous fentanyl will be administered for the procedural pain relief. Post procedural pain relief will be given as deemed necessary by the physician.

Technical success is defined as delivery of all the DEBIRI or when stasis has been reached in the hepatic artery.

Patients will be expected to stay in the hospital for at least a day for monitoring of adverse events, after which they will be followed up in the clinic.

Procedures will be delayed at the physician's discretion should:

* Liver function tests and bilirubin 5-folds more than the normal values
* Absolute neutrophil count of less than 1500 cells/µL
* Platelet count of less than 100,000/µL
* Severe adverse events.

Should the patient development significant extrahepatic metastases at any time during the course of the trial, the referring clinician may choose to stop the trial and/or offer patients other treatment modalities e.g. radiotherapy or further lines of chemotherapy.

4)Follow up:

Patients will be expected to stay in the hospital for at least a day for monitoring of adverse events, after which they will be followed up in the clinic. All patients will be seen in the clinical 1 week after each procedure with FBC and LFT determinations being performed. They will then be seen in the clinic 1 week prior to their next procedure.

Patients will be followed up 3 months after the last procedure. Serum drug levels and adverse events will be monitored. Imaging response will be determined by modified RECIST criteria.

A CT scan will be performed 1 month and 3 months after completion of the procedure to evaluate treatment response. Tumor response will be determined using modified RECIST criteria (7).

5)Pharmacokinetics of irinotecan Blood samples (3 mL) for pharmacokinetic analyses will be collected at the following time points after administration of the first dose on day 1: 0 minutes (pretreatment blank), 1h, 2h, 4h, 8h and 24h hours postinfusion. Blood will be immediately centrifuged at 2000 g for fifteen minutes, and the plasma transferred to a 1.5 mL polypropylene tube and stored at -20°C. Irinotecan and its metabolites, SN-38 and SN-38G will be assayed using LC-MS/MS method. The purpose of performing pharmacokinetics would be to quantitate the AUC of irinotecan, SN-38 and SN-38G in plasma.

6)Pharmacogenetics Analysis Pharmacogenetic analyses for UGT1A1*28 and UGT1A1*6 will be done in all patients prior to administration of irinotecan in accordance with previously published studies by our laboratory (6-9). All participating patients will have venous blood samples (3 mL) drawn for genomic DNA collection in EDTA tubes and labeled with the patient's identification number, date of collection, age, ethnic group and sex.

Unused DNA samples from patients enrolled in the genotyping arm will be stored at -20°C for future pharmacogenetic investigations related to irinotecan research. Patients will be informed and written consent will be taken from them.

8)Potential Risks and benefits

Anticipated benefits:

1. Reduction in the size of the liver lesions hence prolonging survival
2. Meeting criteria for liver resection for metastases

Possible risks:

Adverse events related to procedure include:

1. Access site injuries
2. Hepatic artery injury
3. Non target embolization resulting in acute cholecystitis, peptic ulcer, pancreatitis etc.
4. Post embolization syndrome, manifested by fever, malaise, right upper quadrant pain, nausea, and vomiting
5. Hepatic abscess and biloma
6. Biliary strictures
7. Liver failure

Adverse events related to irinotecan include:

1. Diarrhea
2. Vomiting
3. Leucopenia
4. Anemia
5. Thrombocytopenia

7. Abdominal pain 8. Fever

All chemotherapeutic toxicities will be graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC version 3).

Hematological Dose Limiting Toxicity (DLT) is defined as follows: grade 4 neutropenia of >7 days duration, neutropenic fever, grade 4 anemia or grade 3-4 thrombocytopenia that occurs during the first cycle of treatment.

9)Adverse events

Using Health Science Authority's Safety Reporting for Clinical Trials (June 2011), a serious adverse event (experience) or reaction is any untoward medical occurrence that at any dose

1. Results in death
2. Is life-threatening
3. Requires inpatient hospitalisation or prolongation of existing hospitalization
4. Results in persistent or significant disability/incapacity, or
5. A congenital anomaly/birth defect.

An adverse event is defined as: Any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.

Adverse events related to procedure include:

1. Access site injuries
2. Hepatic artery injury
3. Non target embolization resulting in acute cholecystitis, peptic ulcer, pancreatitis etc.
4. Post embolization syndrome, manifested by fever, malaise, right upper quadrant pain, nausea, and vomiting
5. Hepatic abscess and biloma
6. Biliary strictures
7. Liver failure

All chemotherapeutic toxicities will be graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC version 3).

Hematological Dose Limiting Toxicity (DLT) is defined as follows: grade 4 neutropenia of >7 days duration, neutropenic fever, grade 4 anemia or grade 3-4 thrombocytopenia that occurs during the first cycle of treatment.

Non-hematologic DLT is defined as any grade 3 or grade 4 non-hematologic toxicity that occurs during the first cycle of treatment.

Toxicities will be classified as related to the study drug unless they were attributable to either underlying tumour progression, concurrent medical condition or a concomitant medication. Any unusual toxicities must be reported to the Principal Investigator.

10)Safety Monitoring Plan

Data monitoring

- The principle and co-investigators.

Safety monitoring

* The medical practitioner performing the procedure will be overall responsible for the patient prior to, during and after the intervention.
* The monitoring nurse in the recovery area and the circulating nurse during the procedure will assist the medical practitioner in recording and monitoring the patient's parameters.
* All complications and adverse events will be recorded in the CRFs and the patient will be followed up.

In the event of any SAE's regardless of the causality of the event, the investigator will notify to the IRB of SingHealth. The reporting timelines are:

Urgent Reporting: All problems involving local deaths should be reported immediately within 24 hours after first knowledge by the investigator.

Expedited Reporting: All other SAE must be reported as soon as possible but not later than 7 calendar days after first knowledge by the investigator.

A Data & Safety Monitoring Committee (DSMC) comprising of co-principal investigators from the participating centres, will monitor the safety data .

If the DSMC have any safety concerns, they may make written recommendations to the primary PI and the IRB of SingHealth to modify or terminate the study following discussions with the primary PI. The final decision on the termination of the study will be made by SGH after consulting with IRB and HSA about the safety findings or concerns.

11)Confidentiality of Data and Patient Records

Data required according to the protocol will be recorded on the CRFs as soon as possible.

* Entries must be made with a ballpoint pen and written legibly. No pencils or correction fluids will be used.
* Relevant information will be documented into the patient's hospital files (either paper or electronic records).
* Necessary corrections will be entered by the investigator or, if appropriate, by an authorized member of the investigator's staff in the following manner: The wrong entry will be crossed out, although it must remain legible, and the correct entry will be placed next to it. All corrections will be initialed and dated. For corrections concerning adverse events or the primary variable, a reason for any alteration must be provided.
* Any documents related to the study must be archived at the study site or in a central archive. This includes the careful listing of the identities of the patients involved in the study. This list and the signed informed consent statements are key documents in the files to be stored by the investigator.
* Patient (hospital) files will be archived according to local regulations. All documents related to the study must be retained until at least 15 years after the end of the study. At the end of this period, the investigator is to obtain permission from the relevant authorities (IRB) before any documents are destroyed.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic colorectal carcinoma to the liver, both unilobar and bilobar disease
2. Refractory to 1st or 2nd line systemic chemotherapy. Previous chemotherapy had to be discontinued at least 4 weeks prior to study entry
3. Hepatic disease should be 80% or more of total body tumor burden
4. Measurable liver tumour burden was of no more than 60% of the total liver volume.
5. A performance status of 0-2 (WHO criteria).
6. Age <85 years were required.
7. Life expectancy of greater than 3 months
8. Adequate hematologic function (granulocyte count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, INR ≤ 1.3 in patients on anticoagulant therapy)Adequate hepatic function (total bilirubin ≤ 1.5 x the upper limits of normal [ULN], AST and ALT ≤ 5 x ULN, and alkaline phosphatases < 5 x ULN) and,
9. Adequate renal function (creatinine clearance > 50 mL/min)

Exclusion Criteria:

1. Extrahepatic tumor burden of > 20%.
2. Patients with unilobar disease who are candidates for surgical resection.
3. Extensive tumor involvement of the liver (>60%)
4. Poor performance status (>2 WHO criteria)
5. Significant diseases of cardiac, renal, bone marrow or pulmonary apparatus, central nervous system involvement, and uncontrolled infection
6. Liver function tests and bilirubin 5-folds more than the normal value
7. History of other cancer except adequately treated in situ carcinoma of the cervix or basal or squamous carcinoma of the skin
8. Absolute neutrophil count of less than 1500 cells/µL
9. Platelet count of less than 100,000/µL
10. Significant portal vein thrombosis
11. Unable to understand nature of study and provide written consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Establish safety and toxicity profile of the irinotecan loaded DEBIRI beads (number of patients with adverse events according to Health Science Authority's Safety Reporting for Clinical Trials) | 1 year
  By looking at the number of patients with adverse events according to Health Science Authority's Safety Reporting for Clinical Trials (June 2011)

SECONDARY OUTCOMES:
Tumour response (measured by mRECIST) | 6 months
  measured by mRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Kiang Hiong Tay, MBBS FRCR, Principal Investigator — Singapore General Hospital
Locations (2):
- Singapore (2):
  - National Cancer Centre Singapore, Singapore, Singapore
  - Singapore General Hospital, Singapore